CLINICAL TRIAL: NCT04456894
Title: Importance of Monitoring Primary Hemostasis Pathology in Patients on Extracorporeal Membrane Oxygenation (ECMO) During Lung Transplantation
Brief Title: Primary Hemostasis Pathology in Patients on ECMO During Lung Transplantation
Status: Completed | Type: Observational
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Durila Miroslav MUDr. Ph.D., assoc.prof. MD. Miroslav Durila, PhD., University Hospital, Motol
Other Study IDs: 01072020
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: ECMO Primary Hemostasis Pathology
Keywords: ECMO; PFA 200; ROTEMplatelets; bleeding
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Lung transplantation is a very long and difficult procedure accompanied by a number of possible complications. In the vast majority of cases, the operation itself is performed using the ECMO support, which can negatively affect blood clotting, especially the formation of a platelet blood clot, i.e. primary hemostasis. Thus, the procedure may be accompanied by considerable blood loss, which amount can subsequently negatively affect the postoperative period. It can be assumed, that precise diagnosis of primary hemostasis disorders and subsequent targeted therapy can reduce blood loss and improve outcome of the patient. However, the role of primary hemostasis has not yet been sufficiently specified in this area. Usually, coagulation functions during surgery, are at our department monitored by using ROTEM tests (assesses clot strength), PFA 200 (assesses primary haemostasis under high shear stress conditions and is very sensitive to vWF deficiency) and ROTEM / platelet (assesses primary haemostasis under "low shear stress" conditions and is very susceptible to platelet dysfunction). Targeted therapy by administering necessary clotting factors is used, if any pathology in these tests is detected. However, it is not known, whether the targeted therapy administered is effective enough in patients during the support of extracorporeal circulation. In our monocentric, prospective, observational study, data from the tests mentioned above will be analyzed, and their correlation with a laboratory examination of VWF levels and activity will be monitored. Based on these data, we will try to determine whether perioperative examination of primary hemostasis during lung transplantation (PFA examination, Rotem / platelet-aggregometry and von Willebrand factor-vWF level) is of clinical significance and whether the diagnosis of hemostasis disorder at this level and subsequent targeted therapy may reduce perioperative blood loss.

DETAILED DESCRIPTION:
ECMO is a type of extracorporeal circulation that has experienced a significant increase in use in the last decade as a substitute for lung or heart functions in patients, both perioperatively - especially extensive thoracic surgery procedures such as lung transplantation, or in resuscitation care - in life-threatening conditions associated with heart or lung failure. It uses the classical principle of extracorporeal circulation technology to create continuous, non-pulsating blood flow and, at the same time, its extracorporeal oxygenation. In its two basic configurations, it can only be used to provide respiratory support (veno-venous configuration, VV ECMO), or also cardiac support (veno-arterial configuration, VA ECMO).

Due to the fact that ECMO circuit is an artificial system consisting of cannulas, blood pump and oxygenator itself, the blood is exposed to a huge surface that is not covered by endothelium, thus stimulates the activation of proinflammatory and procoagulant systems. This exposure results in a prothrombotic condition that is associated with a high risk of thrombotic complications. At the same time, however, with this continuous activation of the coagulation cascade, platelets and coagulation factors are depleted, this may lead to an increased risk of bleeding. Pathological shear stress may result in direct binding of VWF (von Willebrand factor) and the platelet GPIIb / IIIa receptor, resulting in their activation and thrombotic complications, however, the effect of non-physiological shear stress may also lead to loss of GPIbα and GPVI platelet receptors, which, in the opposite, causes a disorder of their adhesion and aggregation to VWF and collagen and increases risk of bleeding. Another important factor is loss and fragmentation of the large VWF multimers, a condition known as acquired von Willebrand's syndrome, which causes platelet adhesion to be impaired and thus contributes to bleeding complications.

Both of these situations, definitely, increase morbidity and mortality in patients, so it is necessary to find an optimal and reliable options for the coagulation system functions monitoration, based on which it is possible to immediately perform a targeted therapeutic intervention.

Results of several studies suggest, that increased platelet activation or decreased function results in both thrombotic and bleeding complications in patients requiring extracorporeal support, and these changes cannot be detected by tests, which are usually performed (ROTEM or other common coagulation tests).

Hypothesis:

ECMO causes an early disorder of primary hemostasis, which is detectable by point of care (POC) testing methods PFA 200 and ROTEM / platelet, according to their results, targeted and effective therapy can be applied.

Objectives:

Primary objective is to find out:

* whether ECMO implantation leads to an early failure of primary hemostasis, which can be diagnosed by POC examination - PFA 200, Rotem / platelet-aggregometry and von Willebrand factor levels.
* whether targeted therapy of primary hemostasis disorders (based on the results of POC tests) leads to normalization of these tests results and cessation of bleeding

Secondary objectives:

* to determine the extent of correlation of POC tests of primary hemostasis and laboratory examination of VWF function and quantity
* to clarify the correlation between possible pathological values of these tests and clinically significant bleeding in the patient
* identification of the most reliable method for the assessment of primary hemostasis

Methods:

The group of patients will be represented by patients indicated for implantation of ECMO support during the lung transplantation procedure. ROTEM, PFA 200 and ROTEM / platelet POCs will be used for the perioperative detection of primary and secondary hemostasis disorders- this is a standard approach in Motol University Hospital. In addition to these standard tests, an analysis of the blood sample will also be performed in cooperation with the Institute of hematology and blood transfusion. These tests are represented by quantification of vFW (using quantification of vWF antigen), vFW function test - Ristocetin Cofactor Assay (ex vivo examination of patient's blood plasma, which is depleted of platelets but contains vWF) and Colagen Binding Assay (measures the ability of VWF, especially its large multimers, to bind to collagen).

Blood samples will be taken:

1. after induction into general anesthesia
2. shortly (15-60 minutes) after ECMO initiation
3. shortly (10 minutes) after administration of aimed therapy (vWF or platelets)
4. shortly after ECMO explantation (during admission to the ICU, approximatelly 60 minutes after explantation) An informed consent will be signed with the patient prior to lung transplantation.

Time schedule: 1 year (i.e. 40 patients, on average, about 35 patients undergo lung transplantation per year at our department).

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing elective bilateral lung transplantation on ECMO

Exclusion Criteria:

* patients on dual antiplatelets therapy or patients with vWF disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on waiting list for planned lung transplantation procedure. Patients with COPD, cystic fibrosis, interstitial pulmonary fibrosis, primary pulmonary hypertension
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2020-11-07 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
To find out whether ECMO implantation leads to an early failure of primary hemostasis, which can be diagnosed by POC examination - PFA 200, Rotem / platelet-aggregometry and von Willebrand factor levels | 1 year
  To compare primary hemostasis before and after ECMO implantation
To find out whether targeted therapy of primary hemostasis disorders (based on the results of POC tests) leads to normalization of these tests results and cessation of bleeding | 1 year
  To evaluate whether aimed therapy based on results of POC tests leads to improvement of test results and bleeding
To find out whether aimed treatment during ECMO will be effective or whether primary hemostasis pathology can be by-passed by activated FVIIa | 1 year
  In case that aimed therapy does not stop bleeding or improved POC tests, activated FVIIa in small dose of 15-30 ug/kg can be used to ,,by-pass" primary hemostasis

SECONDARY OUTCOMES:
To determine the extent of correlation of POC tests of primary hemostasis and laboratory examination of VWF function and quantity | 1 year
To identify the most reliable method for the assessment of primary hemostasis | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- UH Motol, Prague, Česká Republika, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garaj M, Durila M, Vajter J, Solcova M, Marecek F, Hrachovinova I. Extracorporeal membrane oxygenation seems to induce impairment of primary hemostasis pathology as measured by a Multiplate analyzer: An observational retrospective study. Artif Organs. 2022 May;46(5):899-907. doi: 10.1111/aor.14142. Epub 2021 Dec 17. PMID 34904233
- [Background] Durila M, Vajter J, Garaj M, Smetak T, Hedvicak P, Berousek J, Vymazal T. Acquired primary hemostasis pathology detected by platelet function analyzer 200 seen during extracorporeal membrane oxygenation is sufficient to prevent circuit thrombosis: A pilot study. J Heart Lung Transplant. 2020 Sep;39(9):980-982. doi: 10.1016/j.healun.2020.05.015. Epub 2020 Jun 11. No abstract available. PMID 32591313
- [Background] Garaj M, Francesconi A, Durila M, Vajter J, Holubova G, Hrachovinova I. ECMO produces very rapid changes in primary hemostasis detected by PFA-200 during lung transplantation: An observational study. J Heart Lung Transplant. 2024 Nov;43(11):1771-1776. doi: 10.1016/j.healun.2024.07.012. Epub 2024 Jul 20. PMID 39038564
- [Background] Lafc G, Budak AB, Yener AU, Cicek OF. Use of extracorporeal membrane oxygenation in adults. Heart Lung Circ. 2014 Jan;23(1):10-23. doi: 10.1016/j.hlc.2013.08.009. Epub 2013 Sep 1. PMID 24144910
- [Background] Hayanga JWA, Chan EG, Musgrove K, Leung A, Shigemura N, Hayanga HK. Extracorporeal Membrane Oxygenation in the Perioperative Care of the Lung Transplant Patient. Semin Cardiothorac Vasc Anesth. 2020 Mar;24(1):45-53. doi: 10.1177/1089253219896123. Epub 2020 Jan 2. PMID 31893982
- [Background] Chen Z, Mondal NK, Ding J, Koenig SC, Slaughter MS, Wu ZJ. Paradoxical Effect of Nonphysiological Shear Stress on Platelets and von Willebrand Factor. Artif Organs. 2016 Jul;40(7):659-68. doi: 10.1111/aor.12606. Epub 2015 Nov 18. PMID 26582038
- [Background] Balle CM, Jeppesen AN, Christensen S, Hvas AM. Platelet Function During Extracorporeal Membrane Oxygenation in Adult Patients. Front Cardiovasc Med. 2019 Aug 8;6:114. doi: 10.3389/fcvm.2019.00114. eCollection 2019. PMID 31440518
- [Background] Heilmann C, Geisen U, Beyersdorf F, Nakamura L, Benk C, Trummer G, Berchtold-Herz M, Schlensak C, Zieger B. Acquired von Willebrand syndrome in patients with extracorporeal life support (ECLS). Intensive Care Med. 2012 Jan;38(1):62-8. doi: 10.1007/s00134-011-2370-6. Epub 2011 Oct 1. PMID 21965100
- [Background] Chen Z, Mondal NK, Zheng S, Koenig SC, Slaughter MS, Griffith BP, Wu ZJ. High shear induces platelet dysfunction leading to enhanced thrombotic propensity and diminished hemostatic capacity. Platelets. 2019;30(1):112-119. doi: 10.1080/09537104.2017.1384542. Epub 2017 Nov 28. PMID 29182470
- [Background] Favaloro EJ. Clinical utility of the PFA-100. Semin Thromb Hemost. 2008 Nov;34(8):709-33. doi: 10.1055/s-0029-1145254. Epub 2009 Feb 12. PMID 19214910